CLINICAL TRIAL: NCT02824172
Title: Treatment of the Osgood Schlatter Disease by Immobilization ( Ankle Cruro Resin ) Versus Sporting Rest ( Reference Treatment ) : Randomized Controlled Study
Brief Title: Treatment of the Osgood Schlatter
Acronym: OSGOOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL16_0404
Record Dates: First submitted 2016-06-29; First posted 2016-07-06 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Osgood Schlatter Disease
Keywords: Cast immobilization; Complete rest; Osgood Schlatter
MeSH Terms: conditions — Osteochondrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cast immobilization (Experimental): 36 patients in the experimental cast immobilization
  Interventions: Other: cast immobilization group
- complete sport rest (Active Comparator): 36 patients in the complete sport rest group
  Interventions: Other: complete sport rest.

INTERVENTIONS:
Other: cast immobilization group — Patients in this group will have their knee locked with a resin going from the ankle to the top of the thigh for 4 weeks, followed by 4 weeks without cast but with rehabilitation through physiotherapy.
  Arms: Cast immobilization
Other: complete sport rest. — Patients included in this group will follow the current standard procedure for this disease that is to say complete sport rest during 8 weeks including rehabilitation through physiotherapy, following the exact same technic as the experimental group .
  Arms: complete sport rest

SUMMARY:
The disease Osgood-Schlatter is most commonly found in sports teenager growing up apophysose accounting for 28.4% of osteochondrosis by Breck. It relates to 62% of osteochondrosis knee and affects adolescent girls between 10 and 12 and boys between 12 and 15 It is usually considered a benign pathology that cures in the majority of cases. However, in 5-10% of cases there is persistent residual pain in adulthood.

The classic complication is the avulsion fracture of the tibial tuberosity in adolescents who continued his sports without restriction.

The possible consequences are numerous including the presence of a free bone fragment at the insertion of the tendon originally described by Osgood the establishment of a genu recurvatum, a high kneecap or patella alta and an enlarged tibial tuberosity (ATT) annoying sport.

The main two treatments are complete rest from sport activity or cast immobilization.

The main objective is to compare these two technics according to the proportion of full sporting recovering at 12 months

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls
* From 9 to 15 years old
* Coming to consult in the Sports' medicine ward
* Patients diagnosed with Osgood-Schlatter disease defined by a swelling of the anterior tibial tuberosity (ATT) , pain on palpation of the ATT , pain with passive knee flexion , pain thwarted knee extension and soft rays in profile knee radiography according to the classification of Woolfrey and Chandler (types A -C
* Unilateral or bilateral
* Previously treated or not
* Agreed to participate
* Agreement of the parents to participate
* Affiliation to national security

Exclusion Criteria:

* Contraindication to the set-up of vascular access in femoral position (femoral Scarpa wound, aortic dissection)
* Local infection
* Hypothermia <32°C
* Need for implementation of arterial catheter only
* Need for implementation of venous catheter only

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Restarting a sporting activity | 12 weeks after intervention
  Comparison between the 2 groups of the proportion of patient returning to sports activity 12 weeks after treatment.

SECONDARY OUTCOMES:
Anterior tibial tuberosity pain | Inclusion visit Day 0
  Mean pain evaluation using Visual analogic scale between the 2 groups, at Anterior tibial tuberosity palpation
Anterior tibial tuberosity pain | follow-up visit week 4
  Mean pain evaluation using Visual analogic scale between the 2 groups, at Anterior tibial tuberosity palpation
Anterior tibial tuberosity pain | follow-up visit week 8
  Mean pain evaluation using Visual analogic scale between the 2 groups, at Anterior tibial tuberosity palpation
Anterior tibial tuberosity pain | follow-up visit week 12
  Mean pain evaluation using Visual analogic scale between the 2 groups, at Anterior tibial tuberosity palpation
Pain killer consumption | follow-up visit week 4
  Evaluation of pain killer consumption (type, dose ,frequency) between the 2 groups
Pain killer consumption | follow-up visit week 8
  Evaluation of pain killer consumption (type, dose ,frequency) between the 2 groups
Quality of life assessment | inclusion visit Day 0
  Quality of life will be assessed using the SF-12 auto questionnaire
Quality of life assessment | follow-up visit week 12
  Quality of life will be assessed using the SF-12 auto questionnaire
Quality of life assessment | follow-up visit month 6
  Quality of life will be assessed using the SF-12 auto questionnaire. As the standard follow-up visit are over, this questionnaire will be asked by phone
Activity level assessment | inclusion visit Day 0
  Activity level will be assessed using the Tegner scale
Activity level assessment | follow-up visit week 12
  Activity level will be assessed using the Tegner scale
Activity level assessment | follow-up visit month 6
  Activity level will be assessed using the Tegner scale. As the standard follow-up visit are over, this scale will be asked by phone
complete sport rest compliance assessment | follow-up visit week 4
  The complete sport rest compliance will be assessed using a visual analogic scale (0 to 10, 0 will be a complete rest compliance)
painfulness due to immobilization cast | follow-up visit week 12
  The patient in the cast immobilization group will be asked what was the level his/her level of cast tolerance: bad, average, good or very good.
Quadricipital shortness | inclusion visit Day 0
  The Quadricipital shortness will be evaluated thanks to the knee flexion angle will be measured using the modified Thomas test as well as hamstring muscles length measured using the popliteal angle
Quadricipital shortness | follow-up visit week 4
  The Quadricipital shortness will be evaluated thanks to the knee flexion angle will be measured using the modified Thomas test as well as hamstring muscles length measured using the popliteal angle
Quadricipital shortness | follow-up visit week 8
  The Quadricipital shortness will be evaluated thanks to the knee flexion angle will be measured using the modified Thomas test as well as hamstring muscles length measured using the popliteal angle
Patella size | inclusion visit Day 0
  The patella size will be measure on the lateral radiograph using the Caton and Deschamp index
Patella size | follow-up visit week 8
  The patella size will be measure on the lateral radiograph using the Caton and Deschamp index
Radiographic evolution of Osgood Schlatter disease | follow-up visit week 12
  Both clinicians and radiologist will evaluate separately the evolution of Osgood Schlatter disease using a new classification. It is based on 3 parameters: anterior tibial tuberosity fragmentation, thickening of soft tissues and presence or not of an ossicle.
Potential return to sport activity | follow visit week 8
  After a week of training, patients of each group will be evaluated and the clinician will consider the possibility of a potential return to sport activity the week 8 of follow-up
Return to sport activity at the initial level | follow visit month 6
  Six months after the intervention, patients will be called to evaluate if they were able to return to a sport activity at the same level they were before the disease. This proportion will be compared in between both groups
alternative options during the study | follow visit month 6
  Each patient will be ask during the phone interview at 6 months if the consulted another physicians or if they used an alternative to that proposed in our study.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Francois LUCCIANI, MD, Principal Investigator — Department of Sport's medicine, Hospital Edouard Herriot- Hospices Civils de Lyon
Locations (1):
- Department of Sport's medicine, Hospital Edouard Herriot- Hospices Civils de Lyon, 5 Place d'Arsonval, Lyon, France

REFERENCES:
- [Result] Duperron L., Haquin A., Berthiller J., Chotel F., Pialat J-B., Luciani J-F. Étude d'une cohorte de 30 patients immobilisés avec une résine cruro-malléolaire pour une maladie d'Osgood-Schlatter. Science & Sports. 2016;31(6):323-335. doi:10.1016/j.scispo.2016.04.014.